CLINICAL TRIAL: NCT06694441
Title: Noradrenergic Dysregulation, Sleep and Cognition in Older Adults with Insomnia
Acronym: NASC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Daniela Grimaldi, Associate Professor of Neurology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00219832; R01AG081520-01A1 (NIH)
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Insomnia
Keywords: Insomnia; Older Adults; Noradrenergic dysregulation; sleep; cognition; cognitive function
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention on Subjects with Insomnia (Experimental): The intervention in this study will involve 28 (+4) days of daily exposure to bright light (BL) for two 60-minute sessions (morning and afternoon).
  For the intervention, we will use Re-Timer® light glasses emitting light with an intensity of 230μW/cm2 (~500lux) with a green blue 500nm dominant wavelength (between 480-520nm). Light with these characteristics has been shown effective in suppressing melatonin levels supporting their potential to exert effects on other biological non-visual functions associated with exposure to light relevant for this study.
  Throughout the intervention, participants will keep a diary to monitor daily use of the glasses. Participants will have weekly phone calls with the research team to encourage compliance and monitor potential side effects.
  Interventions: Other: Light Exposure
- Dim Red Light (Active Comparator): Participants randomized to the control group will wear for two 60-minute sessions (morning and afternoon) customized dim-red light (RL) control Re-Timer® light glasses (wavelength peak at 632nm, light intensity < 3 lux). Participants will be instructed to wear the light glasses in habitual indoor environments, without engaging in strenuous activities. Throughout the intervention, participants will keep a diary to monitor daily use of the glasses. Participants will have weekly phone calls with the research team to encourage compliance and monitor potential side effects.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Light Exposure — The intervention in this study will involve 28 (+4) days of daily exposure to bright light (BL) for two 60-minute sessions (morning and afternoon). For the intervention, we will use Re-Timer® light glasses emitting light with an intensity of 230μW/cm2 (~500lux) with a green blue 500nm dominant wavelength (between 480-520nm). Light with these characteristics has been shown effective in suppressing melatonin levels supporting their potential to exert effects on other biological non-visual functions associated with exposure to light relevant for this study. Throughout the intervention, participants will keep a diary to monitor daily use of the glasses. Participants will have weekly phone calls with the research team to encourage compliance and monitor potential side effects.
  Arms: Intervention on Subjects with Insomnia
Other: Placebo — Participants randomized to the control group will wear for two 60-minute sessions (morning and afternoon) customized dim-red light (RL) control Re-Timer® light glasses (wavelength peak at 632nm, light intensity < 3 lux).
  Arms: Dim Red Light

SUMMARY:
This study investigates the relationship between the noradrenergic (NA) system, sleep quality, and cognitive function in older adults with insomnia - a population at elevated risk for Alzheimer's disease-related dementias (ADRD) - compared to age and sex matched controls with normal sleep. The study characterizes NA function through multiple approaches: measuring 24-hour plasma levels of norepinephrine (NE) and its brain metabolite 3-methoxy-4-hydroxyphenylglycol (MHPG); evaluating central NA system response using the clonidine suppression test (a presynaptic α2 adrenoreceptor agonist that reduces locus coeruleus NA activity; and employing pupillometry as a non-invasive marker of autonomic function. To explore NA function's mechanistic role in insomnia, the study uses an intervention with bright light exposure to enhance daytime NA activity, with the goal of improving both sleep quality and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 55 years;
2. Independent in activities of daily living and without clinically significant cognitive impairment as determined by a mini-mental status examination (MMSE) score ≥ 26;
3. Due to the effect of reproductive hormones on autonomic regulation, sleep and cognition, women will be postmenopausal;
4. time spent in bed not greater than 8.5 hours;
5. Sedentary, defined as participation in exercise of moderate intensity for less than 30 minutes per day and less than two times per week on a regular basis.
6. average daily light exposure indicative of indoor environments (from questionnaire).

Inclusion criteria for the insomnia group:

1. Meet criteria for chronic insomnia disorder according to the International Classification of Sleep Disorders (3rd Ed.);
2. Subjective sleep efficiency less than 80% and/or awakening earlier than desired if before 6 AM for ≥3 nights/week in the previous 4 weeks;
3. Subjective WASO (sWASO) ≥ 60 minutes for ≥3 nights/week in previous 4 weeks. sWASO will include time spent awake after sleep onset before final awakening + time spent awake in bed attempting to sleep after the final awakening;
4. global PSQI score greater than 5;
5. average daily light exposure indicative of indoor environments (from questionnaire).

Inclusion criteria for the control group:

1. No history of chronic or short-term insomnia disorder according to the International Classification of Sleep Disorders (3rd Ed.);
2. Subjective sleep efficiency greater than 80%;
3. Subjective mean total sleep time of 6.5 hours to 8 hours;
4. Habitual bedtime of 9PM-midnight;
5. PSQI score ≤ 5. Participants in the control group will be matched with the insomnia group on sex and age (±3 years).

Exclusion Criteria:

1. Sleep disorders other than insomnia (restless legs syndrome, parasomnias, REM behavior disorder, circadian rhythm sleep-wake disorder, sleep apnea by STOP questionnaire and apnea hypopnea index (AHI) ≥ 15 by home sleep apnea test;
2. habitual bedtime before 9pm or morning awakening before 5am;
3. History of neurological disorders;
4. History of psychiatric disorders;
5. A Beck depression inventory ((BDI-II) score greater than 16);
6. Unstable or serious medical conditions;
7. Diabetes;
8. Current, or use within the past month, of psychoactive, hypnotic, stimulant or analgesic medications (except occasionally);
9. Use of medications that interfere with NA system activity including B-blockers, selective serotonin and norepinephrine reuptake inhibitors (SNRIs) and selective norepinephrine-dopamine reuptake inhibitors (NDRIs);
10. Hormone replacement therapy;
11. Use of medications that affects pupil diameter and responses to light (i.e. antihistamines, anticholinergics, benzodiazepines, narcotics for pain;
12. History of visual abnormalities that may interfere with pupillary responses to light exposure such as significant cataracts, narrow-angle glaucoma or blindness;
13. History of heart conditions (i.e. arrhythmia, coronary artery disease, angina, heart failure);
14. Shift work or other types of self-imposed irregular sleep schedules;
15. BMI > 30 kg/m2;
16. History of habitual smoking (6 or more cigarettes/week) or caffeine consumption > 400 mg/day.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
24h plasma norepinephrine | Enrollment to the end of treatment at 10 weeks.
  24-h plasma norepinephrine (pg/mL) collected every two hours
Clonidine suppression test | Enrollment
  Plasma norepinephrine levels (pg/mL) and 3- plasma 3-methoxy-4-hydroxyphenylglycol (MHPG, ng/mL) levels in response to clonidine suppression test. Collected at baseline and every 30 minutes for 2 hours after clonidine ingestion.
Wake after sleep onset (WASO) | Enrollment to the end of treatment at 10 weeks.
  Duration in minutes obtained from polysomnography and actigraphy
Slow oscillatory activity during sleep | Enrollment to the end of treatment at 10 weeks.
  SO activity (0.5 - 1Hz) is measured from EEG during in laboratory stay
Pittsburg Sleep Quality Index | Enrollment to the end of treatment at 10 weeks.
  Self administered questionnaire to evaluate subjective sleep quality
NIH tool box | Enrollment to the end of treatment at 10 weeks.
  Cognitive battery to assess executive functions, attention, episodic and working memory

SECONDARY OUTCOMES:
24-h plasma 3-methoxy-4-hydroxyphenylglycol (MHPG) | Enrollment to the end of treatment at 10 weeks.
  MHPG (ng/mL) is the main metabolite of Norepinephrine from the brain measured in plasma.
24-h plasma cortisol levels | Enrollment to the end of treatment at 10 weeks.
  24-h plasma cortisol levels (nmol/L) collected every two hours as a measure of autonomic activation
24h plasma melatonin | Enrollment to the end of treatment at 10 weeks.
  24-h plasma melatonin (pg/mL) collected every two hour as a circadian measure
Pupillometry | Enrollment to the end of treatment at 10 weeks.
  Pupil size (measure of autonomic activation)
Psychomotor Vigilance Test | Enrollment to the end of treatment at 10 weeks.
  To assess reaction time (ms)
Wake EEG | Enrollment to the end of treatment at 10 weeks.
  EEG power in alpha band during wake to measure vigilance levels
Heart Rate and Heart Rate Variability | Enrollment to the end of treatment at 10 weeks.
  HR (bpm) and measures of HRV variability (high frequency (HF) component and low frequency to high frequency ratio LF/HF to assess autonomic function and sympatho-vagal balnce
Insomnia Severity Index | Enrollment to the end of treatment at 10 weeks.
  Questionnaire to measure insomnia severity
Visual Analogue Scale | Enrollment to the end of treatment at 10 weeks.
  Scale to measure global vigor ( score 0 to 100) and global alertness (0 to 100). Higher scores indicate greater levels of both vigor and positive affect.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Grimaldi, MD, PhD, Principal Investigator — Northwestern University; Phyllis C Zee, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Center for Circadian and Sleep Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Egroo M, Koshmanova E, Vandewalle G, Jacobs HIL. Importance of the locus coeruleus-norepinephrine system in sleep-wake regulation: Implications for aging and Alzheimer's disease. Sleep Med Rev. 2022 Apr;62:101592. doi: 10.1016/j.smrv.2022.101592. Epub 2022 Jan 21. PMID 35124476
- [Background] Mann DM. The locus coeruleus and its possible role in ageing and degenerative disease of the human central nervous system. Mech Ageing Dev. 1983 Sep;23(1):73-94. doi: 10.1016/0047-6374(83)90100-8. PMID 6228698
- [Background] Cirelli C, Huber R, Gopalakrishnan A, Southard TL, Tononi G. Locus ceruleus control of slow-wave homeostasis. J Neurosci. 2005 May 4;25(18):4503-11. doi: 10.1523/JNEUROSCI.4845-04.2005. PMID 15872097
- [Background] McCrae CS, Rowe MA, Tierney CG, Dautovich ND, Definis AL, McNamara JP. Sleep complaints, subjective and objective sleep patterns, health, psychological adjustment, and daytime functioning in community-dwelling older adults. J Gerontol B Psychol Sci Soc Sci. 2005 Jul;60(4):P182-9. doi: 10.1093/geronb/60.4.p182. PMID 15980285
- [Background] Lim AS, Kowgier M, Yu L, Buchman AS, Bennett DA. Sleep Fragmentation and the Risk of Incident Alzheimer's Disease and Cognitive Decline in Older Persons. Sleep. 2013 Jul 1;36(7):1027-1032. doi: 10.5665/sleep.2802. PMID 23814339
- [Background] Shi L, Chen SJ, Ma MY, Bao YP, Han Y, Wang YM, Shi J, Vitiello MV, Lu L. Sleep disturbances increase the risk of dementia: A systematic review and meta-analysis. Sleep Med Rev. 2018 Aug;40:4-16. doi: 10.1016/j.smrv.2017.06.010. Epub 2017 Jul 6. PMID 28890168
- See also: Center for Circadian and Sleep Medicine Website — https://www.feinberg.northwestern.edu/sleep
- See also: REDCap Initial Screening Eligibility Form — https://redcap.nubic.northwestern.edu/redcap/surveys/?s=WK7CDXRNNTLCWEEK
- Available data/document: Study Overview and Intial Screening Eligibility Form — https://redcap.nubic.northwestern.edu/redcap/surveys/?s=WK7CDXRNNTLCWEEK — Full protocol available via email request: CCSMresearch@northwestern.edu